CLINICAL TRIAL: NCT03269617
Title: PreforPro: A Randomized, Placebo Controlled Crossover Study
Brief Title: PHAGE Study: Bacteriophages as Novel Prebiotics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Collaborators: George Mason University (Other); Metabiomics Corp (Industry)
Responsible Party: Principal Investigator, Tiffany Weir, Associate Professor, Colorado State University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 16-6666HH
Record Dates: First submitted 2017-08-01; First posted 2017-09-01 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Gastrointestinal Disorder, Functional
Keywords: dysbiosis; gut microbiota; bacteriophage; irritable bowel syndrome; gastrointestinal distress; prebiotic
MeSH Terms: conditions — Gastrointestinal Diseases; Dysbiosis; Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: The PHAGE Study is a randomized, double-blind, placebo controlled crossover trial that investigates the utility of four supplemental bacteriophage strains (LH01-Myoviridae, LL5-Siphoviridae, T4D-Myoviridae, and LL12-Myoviridae) to modulate the gut microbiota, and therefore ameliorate common inflammation-related GI distress symptoms (e.g., gas, bloating, diarrhea, constipation, etc) experienced by healthy individuals.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Samples were provided in coded bottles whose identity is known only to the product manufacturer. Blinding will persist until all samples have been processed and the data statistically analyzed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Comparator (Placebo Comparator): Placebo control: 1 capsule containing rice maltodextrin consumed 1x daily for 28 days.
  Interventions: Other: Placebo Control
- Experimental (Experimental): Bacteriophage mixture: 1 capsule containing rice maltodextrin and a mixture of 4 bacteriophages consumed 1x daily for 28 days.
  Interventions: Dietary Supplement: Bacteriophage mixture

INTERVENTIONS:
Dietary Supplement: Bacteriophage mixture — Four bacteriophage strains: LH01-Myoviridae, LL5-Siphoviridae, T4D-Myoviridae, and LL12-Myoviridae.
  Other Names: PreforPro
  Arms: Experimental
Other: Placebo Control — Placebo control capsule consisting of rice maltodextrin
  Other Names: rice maltodextrin
  Arms: Placebo Comparator

SUMMARY:
The PHAGE study is designed to determine if a commercial prebiotic product can change the composition of bacteria in the gut for improved intestinal health. A prebiotic is defined as an indigestible dietary component that selectively enhances specific bacterial species in the intestines to confer a health benefit. In this study, the prebiotic a unique combination of bacteriophages, or viruses that infect bacteria. These phages are generally regarded as safe for human consumption and work by infecting bad bacteria in the gut, which allows beneficial bacteria populations to increase. The product, PreforPro, has shown to be effective in culture-based and animal studies, but its efficacy has not been demonstrated in humans. The goal of this study is to see if PreforPro consumption improves gut bacteria profiles in individuals relative to a placebo control and is associated with reduced incidence and severity of gastrointestinal distress.

DETAILED DESCRIPTION:
The goal of this study is to see if consumption of PreforPro, a commercially available prebiotic dietary supplement consisting of a mixture of bacteriophages, improves gut bacteria profiles in individuals relative to a placebo control. Secondary outcome measures include determining changes in comprehensive metabolic profiles, inflammatory markers (systemic and local), microbial metabolites, and perceptions of gastrointestinal distress. To accomplish these research goals, 40 male and female volunteers between 18-65 years old with BMI scores of 20 to 34.9 who suffer from mild gastrointestinal distress will be enrolled.Recruitment will be by referral from local practitioners and through email solicitations. Eligibility will be determined at the Colorado State University Medical Nutrition Therapy Laboratory (MNTL) by a screening questionnaire and interview/assessment by the clinical coordinator. After determining eligibility and securing consent, participants will randomly be assigned to 1 of 2 treatment groups: prebiotic or placebo. Participants will consume one capsule daily of respective treatments for a period of four (4) weeks. At the beginning and end of the 4 week treatment periods blood and stool samples will be collected at the Human Performance Clinical Research Laboratory (HPCRL). This means that participants will make a total of four (4) clinic visits during each treatment period. Following the initial treatment period, all participants will be required to undergo a wash-out period for two (2) weeks. Upon completion of the wash-out period, participants will switch treatment groups for a period of four (4) weeks. Clinic visits at baseline and 4-weeks for collection of stool and blood samples will also be conducted during the second treatment period. Study participants will be required to provide a total of four (4) fecal samples and four (4) fasting blood samples. Additionally, study participants will be required to provide a weekly assessment of GI symptoms during the two treatment periods. All blood samples will be collected at Colorado State University by trained professionals. Fecal sample collection will be performed by the study participant with collection materials provided by study personnel. Both participants and researchers will be blinded during the course of the intervention and throughout the data analysis period. Blinding will be conducted by individuals from Deerland Enzymes, the company that is providing the capsules for intervention.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults
* 18-65 years old
* Mild to moderate GI distress (self-assessed)

Exclusion Criteria:

* Pregnant or breastfeeding
* Diagnosed GI disease (Celiac, peptic ulcer, ulcerative colitis, Crohn's disease, cancer, or other gastrointestinal or metabolic diseases)
* Antibiotic use in the past 2 months
* Use of NSAIDS, statins, metformin, and other drugs known to modify the gut microbiota
* BMI less than 18.0 or greater than 35.0

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-05-30 (Actual)

PRIMARY OUTCOMES:
Microbiota modulation | Baseline visit prior to starting treatments,4 weeks after starting treatment 1, end of 2-week washout period, 4-weeks after starting treatment 2
  Use of 16s rRNA sequencing of stool samples to determine whether the administered interventions resulted in changes to microbial composition.

SECONDARY OUTCOMES:
Local inflammation | Baseline visit prior to starting treatments,4 weeks after starting treatment 1, end of 2-week washout period, 4-weeks after starting treatment 2
  Inflammation in the bowels will be assessed by use of ELISA test for fecal calprotectin.
Systemic Inflammation | Baseline visit prior to starting treatments,4 weeks after starting treatment 1, end of 2-week washout period, 4-weeks after starting treatment 2
  Systemic inflammation will be assessed by an ELISA test for CRP and circulating cytokines and immune factors.

OTHER OUTCOMES:
Microbial metabolism | Baseline visit prior to starting treatments,4 weeks after starting treatment 1, end of 2-week washout period, 4-weeks after starting treatment 2
  Fermentation by microbes in the gut will be assessed by measuring fecal short chain fatty acid concentrations.
Circulating lipids | Baseline visit prior to starting treatments,4 weeks after starting treatment 1, end of 2-week washout period, 4-weeks after starting treatment 2
  Total cholesterol, LDL, HDL, and triglycerides will be determined in venous blood using a clinical analyzer (Piccolo Xpress).
Comprehensive metabolic panel | Baseline visit prior to starting treatments,4 weeks after starting treatment 1, end of 2-week washout period, 4-weeks after starting treatment 2
  Basic metabolic parameters such as fasting glucose, and levels of BUN, creatinine, and liver enzymes will be determined from a single 200 ul aliquot of venous blood using a CMP clinical analysis panel for Piccolo Xpress.
GI symptom self-assessment | Baseline visit prior to starting treatments,4 weeks after starting treatment 1, end of 2-week washout period, 4-weeks after starting treatment 2
  Participants will complete a validated questionnaire to track changes in GI symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Weir, PhD, Principal Investigator — Colorado State University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Febvre HP, Rao S, Gindin M, Goodwin NDM, Finer E, Vivanco JS, Lu S, Manter DK, Wallace TC, Weir TL. PHAGE Study: Effects of Supplemental Bacteriophage Intake on Inflammation and Gut Microbiota in Healthy Adults. Nutrients. 2019 Mar 20;11(3):666. doi: 10.3390/nu11030666. PMID 30897686
- [Result] Gindin M, Febvre HP, Rao S, Wallace TC, Weir TL. Bacteriophage for Gastrointestinal Health (PHAGE) Study: Evaluating the Safety and Tolerability of Supplemental Bacteriophage Consumption. J Am Coll Nutr. 2019 Jan;38(1):68-75. doi: 10.1080/07315724.2018.1483783. Epub 2018 Aug 29. PMID 30157383